CLINICAL TRIAL: NCT01281202
Title: Vigabatrin for Treatment of Cocaine Dependence: A Phase II Study
Brief Title: Vigabatrin for the Treatment of Cocaine Dependency
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Catalyst Pharmaceuticals, Inc. (Industry)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH); VA Office of Research and Development (U.S. Federal Agency)
Responsible Party: Sponsor
Organization: National Institute on Drug Abuse (NIDA) (NIH)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CPP-01005/CS# 1030 TRANSFERRED; Y1-DA4006 (Other Grant/Funding Number: NIDA/VA CSP #1030)
Record Dates: First submitted 2011-01-20; First posted 2011-01-21 (Estimated); Results first posted 2016-02-23 (Estimated); Last update posted 2016-05-18 (Estimated); Status verified 2016-05

CONDITIONS: Cocaine Addiction; Cocaine Dependence
Keywords: Cocaine; Cocaine Addiction Treatment; Cocaine Treatment; Vigabatrin; CPP-109; Catalyst; National Institute on Drug Abuse
MeSH Terms: conditions — Cocaine-Related Disorders | interventions — Vigabatrin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- CPP-109 Vigabatrin Tablets (Active Comparator): Subjects were evaluated for their compliance with protocol inclusion/exclusion criteria during a -2 to -4 week Screening/Baseline Phase
  During treatment, subjects received 3 CPP-109 Vigabatrin 500 mg Tablets, bid, for 9 weeks
  Subjects were provided with on-site, supervised, standardized, manualized Individual Drug Counseling 1x per week for 9 weeks and the first 4 weeks for the follow-up phase (weeks 10-13)
  Interventions: Drug: Vigabatrin
- Placebo (Placebo Comparator): Subjects were evaluated for their compliance with protocol inclusion/exclusion criteria during a -2 to -4 week Screening/Baseline Phase
  During treatment, subjects received Vigabatrin matching placebo tablets, bid, for 9 weeks
  Subjects were provided with on-site, supervised, standardized, manualized Indivdiual Drug Counseling 1x per week for 9 weeks and the first 4 weeks for the follow-up phase (weeks 10-13)
  Interventions: Drug: Matching Placebo

INTERVENTIONS:
Drug: Vigabatrin — Tablets
  Other Names: CPP-109; GVG; VGB
  Arms: CPP-109 Vigabatrin Tablets
Drug: Matching Placebo — Tablets
  Arms: Placebo

SUMMARY:
The objective of this 26-28 week study is to demonstrate that the rate of cocaine dependent subjects treated with CPP-109 vigabatrin in addition to counseling, who completely stop use of cocaine in the last 2 weeks of the study's Treatment Phase (Weeks 8 and 9) will be higher than seen in subjects treated with placebo in addition to counseling.

DETAILED DESCRIPTION:
The objective of this 26-28 week study is to demonstrate that the rate of cocaine dependent subjects treated with CPP-109 vigabatrin in addition to counseling, who completely stop use of cocaine in the last 2 weeks of the study's Treatment Phase (Weeks 8 and 9) will be higher than seen in subjects treated with placebo in addition to counseling.

There are 3 Phases to this study:

* a 2-4 week Screening/Baseline Phase during which eligibility to be included in the trial will be tested;
* a 9 week Treatment Phase during which subjects will receive CPP-109 or placebo tablets in addition to counseling; and
* a 15 week Follow-up Phase, during the first 4 weeks (Weeks 10-13) of which subjects will continue to receive counseling.

ELIGIBILITY:
Inclusion Criteria:

* Able to understand the study and provide written informed consent.
* Male or female at least 18 years of age.
* Meet DSM-IV criteria for cocaine dependence as primary diagnosis, as determined by the Substance Abuse Structured Clinical Interview (SCID) for Diagnostic and Statistical Manual-IV (DSM-IV) module.
* Have a verifiable place of primary residence.
* Seeking treatment for cocaine dependence.
* Be in generally good health based on history, physical examination, electrocardiogram, eye exam and laboratory findings.
* If female of childbearing potential, use acceptable contraceptive methods (oral contraceptives (the pill), intrauterine device (IUD), contraceptive implants under the skin, contraceptive rings or patches or injections, diaphragms with spermicide, and condoms with spermicide). Surgical sterilization by tubal ligation or hysterectomy is acceptable.

Exclusion Criteria:

* Please contact site for more information

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 207 (Actual)
Dates: Start 2011-01; Primary Completion 2012-10 (Actual); Study Completion 2012-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Kathleen Brady, MD, PhD, Principal Investigator — Medical University of South Carolina; Christopher J Stock, PharmD, Study Chair — George E. Wahlen VA Medical Center
Locations (13):
- United States (13):
  - Matrix Institute on Addictions, Los Angeles, California
  - Friends Research Institute, Torrance, California
  - VA Medical Center, Denver, Colorado
  - University of Miami School of Medicine, Miami, Florida
  - NeuroPsychiatric Research & Practice Assoc., Ltd., Oak Brook, Illinois
  - Mountain Manor Treatment Center @ Baltimore, Baltimore, Maryland
  - Boston University School of Medicine, Boston, Massachusetts
  - Pacific Institute for Research and Evaluation, Albuquerque, New Mexico
  - Western Psychiatric Inst. and Clinic, Pittsburgh, Pennsylvania
  - Medical University of South Carolina, Charleston, South Carolina
  - Pillar Clinical Research, LLC, Dallas, Texas
  - University of Texas Health Science Center at Houston, Houston, Texas
  - George E Wahlen VA Medical Center, Salt Lake City, Utah

IPD SHARING:
Plan to Share IPD: Yes

RESULTS

PARTICIPANT FLOW:
Groups:
- CPP-109 Vigabatrin Tablets: Participants received Vigabatrin 3.0 gm tablet orally once daily for 7 weeks.
- Placebo: Participants received Vigabatrin placebo table orally once daily for 7 weeks.
Period: Overall Study
Arm/Group | CPP-109 Vigabatrin Tablets | Placebo
Started | 103 | 104
Completed | 75 | 68
Not Completed | 28 | 36
Not completed — Adverse Event | 2 | 0
Not completed — Withdrawal by Subject | 2 | 2
Not completed — Protocol Violation | 11 | 10
Not completed — Administrative | 2 | 8
Not completed — Lost to Follow-up | 11 | 13
Not completed — Incarceration | 0 | 3

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | CPP-109 Vigabatrin Tablets | Placebo | Total
Number analyzed (Participants) | 103 | 104 | 207
Age, Continuous [Mean (Standard Deviation); unit: years] | 46.1 (7.5) | 47.2 (7.4) | 46.6 (7.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 29 | 33 | 62
  Male | 74 | 71 | 145
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 17 | 18 | 35
  Not Hispanic or Latino | 84 | 85 | 169
  Unknown or Not Reported | 2 | 1 | 3
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 2 | 2
  Asian | 1 | 0 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 55 | 52 | 107
  White | 39 | 39 | 78
  More than one race | 3 | 3 | 6
  Unknown or Not Reported | 5 | 8 | 13
Region of Enrollment [Number; unit: participants]
  United States | 103 | 104 | 207

OUTCOME MEASURES:

1. Primary Outcome: Abstinence
Description: The number of subjects in each treatment group who are cocaine abstinent during the last 2 weeks of the Treatment Phase (Weeks 8 and 9).
Time Frame: Weeks 8-9
Measure: Number; unit: participants
Groups:
- CPP-109 Vigabatrin Tablets: Subjects were evaluated for their compliance with protocol inclusion/exclusion criteria during a -2 to -4 week Screening/Baseline Phase. During treatment, subjects received 3 CPP-109 Vigabatrin 500 mg Tablets, bid, for 9 weeks.
  Subjects were provided with on-site, supervised, standardized, manualized Individual Drug Counseling 1x per week for 9 weeks and the first 4 weeks for the follow-up phase (weeks 10-13)
- Matching Placebo: Subjects were evaluated for their compliance with protocol inclusion/exclusion criteria during a -2 to -4 week Screening/Baseline Phase. During Treatment, subjects received Vigabatrin matching placebo tablets, bid, for 9 weeks.
  Subjects were provided with on-site, supervised, standardized, manualized Individual Drug Counseling 1x per week for 9 weeks and the first 4 weeks for the follow-up phase (weeks 10-13)
Arm/Group | CPP-109 Vigabatrin Tablets | Matching Placebo
Number analyzed (Participants) | 103 | 104
participants | 5 | 9

2. Secondary Outcome: Number of Participants With Cocaine Use
Time Frame: Week 3 - 9
Measure: Number; unit: participants
Groups:
- CPP-109 Vigabatrin Tablets: Subjects were evaluated for their compliance with protocol inclusion/exclusion criteria during a -2 to -4 week Screening/Baseline Phase
  During treatment, subject received 3 CPP-109 Vigabatrin 500 mg Tablets, bid, for 9 weeks
  Subjects were provided with on-site, supervised, standardized, manualized Individual Drug Counseling 1x per week for 9 weeks and the first 4 weeks for the follow-up phase (weeks 10-13)
- Placebo: Subjects were evaluated for their compliance with protocol inclusion/exclusion criteria during a -2 to -4 week Screening/Baseline Phase
  During treatment, subject received Vigabatrin matching placebo tablets, bid, for 9 weeks
  Subject were provided with on-site, supervised, standardized, manualized Individual Drug Counseling 1x per week for 9 weeks and the first 4 weeks for the follow-up phase (weeks 10-13)
Arm/Group | CPP-109 Vigabatrin Tablets | Placebo
Number analyzed (Participants) | 103 | 104
participants
  Week 3 | 95 | 96
  Week 4 | 91 | 95
  Week 5 | 88 | 93
  Week 6 | 86 | 90
  Week 7 | 84 | 85
  Week 8 | 83 | 82
  Week 9 | 81 | 81

ADVERSE EVENTS:
Arm/Group | CPP-109 Vigabatrin Tablets | Placebo
Serious Adverse Events (participants affected / at risk) | 6/103 | 3/104
Other Adverse Events (participants affected / at risk) | 84/103 | 89/104
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | CPP-109 Vigabatrin Tablets (N=103) | Placebo (N=104)
Chest Pain (General disorders) | 2 | 1
Depression suicidal (Psychiatric disorders) | 0 | 1
Psychiatric symptom (Psychiatric disorders) | 1 | 0
Blood pressure increased (Investigations) | 1 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 1
Loss of conciousness (Nervous system disorders) | 1 | 0
Eczema (Skin and subcutaneous tissue disorders) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | CPP-109 Vigabatrin Tablets (N=103) | Placebo (N=104)
Nausea (Gastrointestinal disorders) | 8 | 25
Headache (Nervous system disorders) | 22 | 29
Back pain (Musculoskeletal and connective tissue disorders) | 8 | 13
Pain in extremity (Musculoskeletal and connective tissue disorders) | 11 | 8
Fatigue (General disorders) | 16 | 13
Insomnia (Psychiatric disorders) | 4 | 8
Nasopharyngitis (Respiratory, thoracic and mediastinal disorders) | 9 | 7
Contusion (Injury, poisoning and procedural complications) | 3 | 8
Photopsia (Eye disorders) | 11 | 2
Blood pressure increased (Investigations) | 8 | 4
Pruritus (Skin and subcutaneous tissue disorders) | 5 | 1
Hypertension (Vascular disorders) | 4 | 14
Dysmenorrhoea (Reproductive system and breast disorders) | 1 | 5
Increased appetite (Metabolism and nutrition disorders) | 4 | 3
Immune system disorders (Renal and urinary disorders) | 4 | 3

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days